CLINICAL TRIAL: NCT02668224
Title: Chronic Effects of Tendon Vibrations on the Neuromechanical Muscular Properties : Pilot Study, Interventional, Prospective, Longitudinal.
Brief Title: Chronic Effects of Tendon Vibrations on the Neuromechanical Muscular Properties.
Acronym: NEUROVIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1408208; 2015-A00036-43 (Other: ANSM)
Record Dates: First submitted 2016-01-22; First posted 2016-01-29 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vibrasens : Test group (Experimental): Training programme: vibration training 3/week from Day 1 to Day 60 + Usual activities from day 60 to Day 75.
  Interventions: Device: Vibrasens
- Control group (Active Comparator): Control: Usual activities from day 1 to Day 75.
  Interventions: Other: Usual activities

INTERVENTIONS:
Device: Vibrasens — Transcutaneous vibrations are used. This device allows vibrations from 25 to 150 Hz with an amplitude of 1 mm. In our study the frequency used is 50 Hz.
  Arms: Vibrasens : Test group
Other: Usual activities — The patients will perform their usual activities, to allow the comparison with a vibration programme. They will not have a specific training.
  Arms: Control group

SUMMARY:
It is a randomized, controlled clinical trial, in healthy volunteers. They are in two groups : the test one will perform the vibration training (1h of Vibrasens 3 times a week, 24 sessions) whereas the control group will not be training. The primary outcome is the maximal voluntary strength.

DETAILED DESCRIPTION:
These last 10 years, a new idea born: vibrations could have potential effects on muscular reconditioning. Researchers have previously demonstrated the effects on plantar ankle flexion, with the increase of the strength, on healthy volunteers. Nowadays physicians would like to demonstrate the effects on another muscular group: ankle's dorsal flexors. 24 sessions are programmed on 8 weeks.

Moreover, the last results showed a modification of the nervous capacities of the cortical voluntary activation. Transcranial Magnetic Stimulation (TMS) is a great tool to explore the neuromuscular function, at the cortical stage. The use of this tool will allow the characterization the effects of the vibration training on the cortical activation state.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years old
* Both gender
* Occasional sportsman (<4h/week)
* Affiliated to a social security scheme
* Having freely given their written consent

Exclusion Criteria:

* Taking neuro-active substances able to modify cortico-spinal excitability from Day 10 to the end of the study
* Contraindication to magnetic field application
* Previous pathologies susceptible to modify the process of the tests (particularly stakeholders presenting knee or ankle pathologies)
* Participation during the same time in another interventional experimentation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Increase of maximal voluntary strength in dorsal flexion of the ankle | 8 weeks
  Determine if a training of 24 sessions of tendon vibrations of dorsal flexors' ankles programmed on 8 weeks allows the increase of the maximal voluntary strength in ankles' dorsal flexion, compared to a control group, with no vibration.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard FEASSON, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No